CLINICAL TRIAL: NCT05972200
Title: Probing the Efficacy of V5/MT Stimulation on Reading and Reading-related Measures in Children and Adolescents With Developmental Dyslexia
Brief Title: V5/MT Stimulation on Reading and Reading-related Measures in Developmental Dyslexia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Deny Menghini, Head of Psychology Unit, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3073_OPBG_2023
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Developmental Dyslexia
Keywords: Children; Adolescents; tDCS; transcranial direct current stimulation; neurodevelopmental disorders; non-invasive brain stimulation; transcranial electrical stimulation; EEG; reading abilities
MeSH Terms: conditions — Dyslexia; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- HD-tDCS V5/MT, HD-tDCS V1, Sham (Experimental): 1. Active HD-tDCS over V5/MT
  2. Active HD-tDCS over V1
  3. Sham HD-tDCS over V5/MT or V1
  Interventions: Device: Active HD-tDCS over V5/MT; Device: Active HD-tDCS over V1; Device: Sham HD-tDCS over V5/MT or V1
- HD-tDCS V5/MT, Sham, HD-tDCS V1 (Experimental): 1. Active HD-tDCS over V5/MT
  2. Sham HD-tDCS over V5/MT or V1
  3. Active HD-tDCS over V1
  Interventions: Device: Active HD-tDCS over V5/MT; Device: Active HD-tDCS over V1; Device: Sham HD-tDCS over V5/MT or V1
- HD-tDCS V1, HD-tDCS V5/MT, Sham (Experimental): 1. Active HD-tDCS over V1
  2. Active HD-tDCS over V5/MT
  3. Sham HD-tDCS over V5/MT or V1
  Interventions: Device: Active HD-tDCS over V5/MT; Device: Active HD-tDCS over V1; Device: Sham HD-tDCS over V5/MT or V1
- HD-tDCS V1, Sham, HD-tDCS V5/MT (Experimental): 1. Active HD-tDCS over V1
  2. Sham HD-tDCS over V5/MT or V1
  3. Active HD-tDCS over V5/MT
  Interventions: Device: Active HD-tDCS over V5/MT; Device: Active HD-tDCS over V1; Device: Sham HD-tDCS over V5/MT or V1
- Sham, HD-tDCS V5/MT, HD-tDCS V1 (Experimental): 1. Sham HD-tDCS over V5/MT or V1
  2. Active HD-tDCS over V5/MT
  3. Active HD-tDCS over V1
  Interventions: Device: Active HD-tDCS over V5/MT; Device: Active HD-tDCS over V1; Device: Sham HD-tDCS over V5/MT or V1
- Sham, HD-tDCS V1, HD-tDCS V5/MT (Experimental): 1. Sham HD-tDCS over V5/MT or V1
  2. Active HD-tDCS over V1
  3. Active HD-tDCS over V5/MT
  Interventions: Device: Active HD-tDCS over V5/MT; Device: Active HD-tDCS over V1; Device: Sham HD-tDCS over V5/MT or V1

INTERVENTIONS:
Device: Active HD-tDCS over V5/MT — For HD-tDCS a 4 × 1 montage (Kessler et al., 2013), small circular electrodes (diameter 1 cm) will be used with the anode placed centrally with a current intensity of 1 mA for a total of 20 minutes (30 s ramp up/down). Hereby, the anodal electrode modulates the excitability of the targeted area left V5/MT, whereas the other 4 electrodes return electrical currents that flow away from that area. V5/MT will be localised via published procedures and electrode's placement will be done according to the 10-20 International EEG 10-20 System for electrode placement.
Device: Active HD-tDCS over V1 — For HD-tDCS a 4 × 1 montage (Kessler et al., 2013), small circular electrodes (diameter 1 cm) will be used with the anode placed centrally with a current intensity of 1 mA for a total of 20 minutes (30 s ramp up/down). Hereby, the anodal electrode modulates the excitability of the targeted area left V1, whereas the other 4 electrodes return electrical currents that flow away from that area. V1 will be localised via published procedures and electrode's placement will be done according to the 10-20 International EEG 10-20 System for electrode placement.
Device: Sham HD-tDCS over V5/MT or V1 — Sham HD-tDCS will be delivered over left V5/MT or left V1. The same electrodes placement as well as the stimulation set-up will be used as in the active stimulation conditions, but the current will be applied for 30 s and will be ramped down (0 mA) during the rest of the session without the participants awareness. .

SUMMARY:
The present study grounds on the absence of evidence-based treatment in individuals with developmental dyslexia (DD). At this topic, the present study will explore the potential effect of transcranial direct current stimulation (tDCS) over left hemispheric direct Lateral Geniculate Nucleus (LGN)-V5/MT pathway, cerebral areas usually disrupted in individuals with DD.

The investigators hypothesized that active tDCS over V5/MT will boost reading skills in children and adolescents with DD. On the contrary, sham (placebo condition) tDCS over V5/MT or active (control condition) tDCS over V1 will not have significant effect in improving reading skills. Further, both active and sham tDCS will be safe and well tolerated.

DETAILED DESCRIPTION:
Over the last few decades, a huge number of studies has revealed that Developmental Dyslexia (DD), a brain-based neurodevelopmental disorder characterized by a severe and persistent impairment in the acquisition of reading skills may depend on multiple neurocognitive impairments, ranging from language-specific to cognitive-general deficits. Besides the most influential hypothesis of a phonological core deficit, there is also evidence for difficulties in low-level visual-temporal information processing, as the magnocellular deficit theory supports, as well as for visual-spatial attentional deficits, visual-perceptual impairments, and rapid automatized naming (RAN)-speed deficits.

Replicated structural/functional neuroimaging studies have demonstrated a DD hypoactivation relative to typical readers in the left temporo-occipital regions-critical for the automatic visual processing of word strings or print-and in the left temporo-parietal regions-important for grapheme-to-phoneme mapping.

Moreover, findings from animal models and post mortem studies in humans suggest that DD might also be associated with structural alterations in subcortical sensory pathways, particularly in visual and auditory thalamic nuclei and in their connections with high-order sensory cortices (i.e., the left hemispheric direct Lateral Geniculate Nucleus (LGN)-V5/MT pathway and the left hemispheric direct Medial Geniculate Body (MGB)-mPT pathway). In addition, in adults with DD, left V5/MT-LGN connectivity strength correlated with RAN abilities - a key deficit in DD.

A number of studies have demonstrated the positive effect of transcranial direct current stimulation (tDCS), a non-invasive brain stimulation used for transiently modifying neural activity of target areas, on reading and, particularly, in DD.

However, the few non-invasive brain stimulation studies on improving reading in DD yielded heterogeneous results and this variability might be partly due to the lack of neurobiological understanding of the underlying DD mechanism or to the use of traditional tDCS rather than a more focal technique such as the high-definition tDCS (HD-tDCS).

Starting from this, the aim of the current study is testing the effectiveness of a cutting-edge stimulation technique (i.e., HD-tDCS) in a within-subject experiment involving children and adolescents with DD. Especially, we will work to test i) the specific effect of HD-tDCS over high-order sensory cortices (i.e., V5/MT vs V1) on reading in children with DD; ii) the preconditions and neurobiological mechanisms that lead to high treatment outcomes.

If the stimulation over V5/MT is effective and specifically related to reading improvement, our results could help to i) understand the contribution and neurobiological mechanism of V5/MT in reading of children and adolescents with DD; ii) select criteria for potential responders to non-invasive brain stimulation; iii) develop evidence-based interventions in DD.

ELIGIBILITY:
Inclusion Criteria:

* Italian speakers right-handed children and adolescents with dyslexia (DSM-5, APA 2013);
* Word/nonword/text reading accuracy and/or speed at least 2 Standard Deviations below the mean for school-age;
* nv IQ ≥ 85;
* normal hearing and normal or corrected-to-normal vision.

Exclusion Criteria:

* Having a comorbidity with other primary psychiatric/neurological diagnosis (e.g., depression, anxiety, autism, ADHD);
* Having a personal history of neurological/medical/genetic diseases;
* Having ongoing drug treatment influencing brain function;
* Having epilepsy o family history of epilepsy.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Text reading accuracy (Experimental reading task) | during procedure
  Change in text reading accuracy from baseline compared after to Active HD-tDCS over V5/MT sessions than after Active HD-tDCS over V1 and Sham sessions. Text reading accuracy is considered as the percentage (%) of accuracy and computed as the ratio between the number of correctly read stimuli and the total number of stimuli presented multiplied by 100.
  The time points will be pre- (baseline) vs post-stimulation session.
Text reading speed (Experimental reading task) | during procedure
  Change in text reading speed from baseline compared to after Active HD-tDCS over V5/MT sessions than after Active HD-tDCS over V1 and Sham sessions. Text reading speed is considered as the syllables/seconds ratio and calculated dividing the total number of syllables pronounced by the total time spent to complete the reading (in seconds).
  The time points will be pre- (baseline) vs post-stimulation session.

SECONDARY OUTCOMES:
Word reading accuracy (Experimental reading task) | during procedure
  Change in word reading accuracy from baseline compared to after Active HD-tDCS over V5/MT sessions than after Active HD-tDCS over V1 and Sham sessions. Word reading accuracy is considered as the percentage (%) of accuracy and computed as the ratio between the number of correctly read stimuli and the total number of stimuli presented multiplied by 100.
  The time points will be pre- (baseline) vs post-stimulation session.
Word reading speed (Experimental reading task) | during procedure
  Change in word reading speed from baseline compared to after Active HD-tDCS over V5/MT sessions than during Active HD-tDCS over V1 and Sham sessions. Word reading speed is considered as the syllables/seconds ratio and calculated dividing the total number of syllables pronounced by the total time spent to complete the reading (in seconds).
  The time points will be pre- (baseline) vs post-stimulation session.
Non-word reading accuracy (Experimental reading task) | during procedure
  Change in non-word reading accuracy from baseline compared to after Active HD-tDCS over V5/MT sessions than after Active HD-tDCS over V1 and Sham sessions. Non-word reading accuracy is considered as the percentage (%) of accuracy and computed as the ratio between the number of correctly read stimuli and the total number of stimuli presented multiplied by 100.
  The time points will be pre- (baseline) vs post-stimulation session.
Non-word reading speed (Experimental reading task) | during procedure
  Change in non-word reading speed from baseline compared to after Active HD-tDCS over V5/MT sessions than after Active HD-tDCS over V1 and Sham sessions. Non-word reading speed is considered as the syllables/seconds ratio and calculated dividing the total number of syllables pronounced by the total time spent to complete the reading (in seconds).
  The time points will be pre- (baseline) vs post-stimulation session.
Right visual hemisphere-motion perception (Experimental reading task) | during procedure
  Change in right visual hemisphere-motion perception from baseline compared to after Active HD-tDCS over V5/MT sessions than after Active HD-tDCS over V1 and Sham sessions. Right visual hemisphere-motion perception is considered as the number of correct saccades.
  The time points will be pre- (baseline) vs post-stimulation session.
Rapid automatized naming letter and number (Experimental reading task) | during procedure
  Change in rapid automatized naming letter and number from baseline compared to after Active HD-tDCS over V5/MT sessions than after Active HD-tDCS over V1 and Sham sessions. Rapid automatized naming letter and number is considered as the total time spent (in seconds) to complete the task.
  The time points will be pre- (baseline) vs post-stimulation session.
Phoneme blending (Experimental reading task) | during procedure
  Change in phoneme blending from baseline compared to after Active HD-tDCS over V5/MT sessions than after Active HD-tDCS over V1 and Sham sessions. Phoneme blending is considered as the number of correctly blended phonemes.
  The time points will be pre- (baseline) vs post-stimulation session.
Eye-movements during reading (Experimental reading task) | during procedure
  Change in eye-movements from baseline compared to after reading during Active HD-tDCS over V5/MT sessions than after Active HD-tDCS over V1 and Sham sessions. Eye-movements during reading is considered as the number of saccades and the number of dwells.
  The time points will be pre- (baseline) vs post-stimulation session.
Spontaneous EEG (Experimental reading task) | during procedure
  Change in spontaneous EEG from baseline compared to after Active HD-tDCS over V5/MT sessions than after Active HD-tDCS over V1 and Sham sessions. Spontaneous EEG is considered as the individual alpha-peak frequency and the beta and theta/gamma oscillations.
  The time points will be pre- (baseline) vs post-stimulation session.

CONTACTS AND LOCATIONS:
Locations (1):
- Bambino Gesù Hospital and Research Institute, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders (5th ed.): DSM 5. Washington, DC: American Psychiatric Association. 2013.
- [Background] Snowling, M. Dyslexia, 2nd ed.; Blackwell Publishing: Oxford, UK. 2000.
- [Background] Wolf M, Bowers PG. The double-deficit hypothesis for the developmental dyslexias. Journal of Educational Psychology. 1999; 91(3): 415-438.
- [Result] Menghini D, Finzi A, Benassi M, Bolzani R, Facoetti A, Giovagnoli S, Ruffino M, Vicari S. Different underlying neurocognitive deficits in developmental dyslexia: a comparative study. Neuropsychologia. 2010 Mar;48(4):863-72. doi: 10.1016/j.neuropsychologia.2009.11.003. Epub 2009 Nov 10. PMID 19909762
- [Result] Vellutino FR, Fletcher JM, Snowling MJ, Scanlon DM. Specific reading disability (dyslexia): what have we learned in the past four decades? J Child Psychol Psychiatry. 2004 Jan;45(1):2-40. doi: 10.1046/j.0021-9630.2003.00305.x. PMID 14959801
- [Result] Melby-Lervag M, Lyster SA, Hulme C. Phonological skills and their role in learning to read: a meta-analytic review. Psychol Bull. 2012 Mar;138(2):322-52. doi: 10.1037/a0026744. Epub 2012 Jan 16. PMID 22250824
- [Result] Schulte-Korne G, Bruder J. Clinical neurophysiology of visual and auditory processing in dyslexia: a review. Clin Neurophysiol. 2010 Nov;121(11):1794-809. doi: 10.1016/j.clinph.2010.04.028. Epub 2010 May 31. PMID 20570212
- [Result] Vidyasagar TR, Pammer K. Dyslexia: a deficit in visuo-spatial attention, not in phonological processing. Trends Cogn Sci. 2010 Feb;14(2):57-63. doi: 10.1016/j.tics.2009.12.003. Epub 2010 Jan 14. PMID 20080053
- [Result] Franceschini S, Gori S, Ruffino M, Pedrolli K, Facoetti A. A causal link between visual spatial attention and reading acquisition. Curr Biol. 2012 May 8;22(9):814-9. doi: 10.1016/j.cub.2012.03.013. Epub 2012 Apr 5. PMID 22483940
- [Result] Bosse ML, Tainturier MJ, Valdois S. Developmental dyslexia: the visual attention span deficit hypothesis. Cognition. 2007 Aug;104(2):198-230. doi: 10.1016/j.cognition.2006.05.009. Epub 2006 Jul 21. PMID 16859667
- [Result] Stenneken P, Egetemeir J, Schulte-Korne G, Muller HJ, Schneider WX, Finke K. Slow perceptual processing at the core of developmental dyslexia: a parameter-based assessment of visual attention. Neuropsychologia. 2011 Oct;49(12):3454-65. doi: 10.1016/j.neuropsychologia.2011.08.021. Epub 2011 Aug 31. PMID 21903119
- [Result] Giovagnoli G, Vicari S, Tomassetti S, Menghini D. The Role of Visual-Spatial Abilities in Dyslexia: Age Differences in Children's Reading? Front Psychol. 2016 Dec 21;7:1997. doi: 10.3389/fpsyg.2016.01997. eCollection 2016. PMID 28066311
- [Result] Wang Z, Cheng-Lai A, Song Y, Cutting L, Jiang Y, Lin O, Meng X, Zhou X. A perceptual learning deficit in Chinese developmental dyslexia as revealed by visual texture discrimination training. Dyslexia. 2014 Aug;20(3):280-96. doi: 10.1002/dys.1475. Epub 2014 Mar 18. PMID 24643918
- [Result] Bowers PG, Wolf, M. Theoretical links among naming speed, precise timing mechanisms and orthographic skill in dyslexia. Reading and Writing.1993; 51: 69-85.
- [Result] Richlan F, Kronbichler M, Wimmer H. Meta-analyzing brain dysfunctions in dyslexic children and adults. Neuroimage. 2011 Jun 1;56(3):1735-42. doi: 10.1016/j.neuroimage.2011.02.040. Epub 2011 Feb 19. PMID 21338695
- [Result] Richlan F. Developmental dyslexia: dysfunction of a left hemisphere reading network. Front Hum Neurosci. 2012 May 1;6:120. doi: 10.3389/fnhum.2012.00120. eCollection 2012. PMID 22557962
- [Result] Livingstone MS, Rosen GD, Drislane FW, Galaburda AM. Physiological and anatomical evidence for a magnocellular defect in developmental dyslexia. Proc Natl Acad Sci U S A. 1991 Sep 15;88(18):7943-7. doi: 10.1073/pnas.88.18.7943. PMID 1896444
- [Result] Galaburda AM, Menard MT, Rosen GD. Evidence for aberrant auditory anatomy in developmental dyslexia. Proc Natl Acad Sci U S A. 1994 Aug 16;91(17):8010-3. doi: 10.1073/pnas.91.17.8010. PMID 8058748
- [Result] Giraldo-Chica M, Hegarty JP 2nd, Schneider KA. Morphological differences in the lateral geniculate nucleus associated with dyslexia. Neuroimage Clin. 2015 Mar 20;7:830-6. doi: 10.1016/j.nicl.2015.03.011. eCollection 2015. PMID 26082892
- [Result] Muller-Axt C, Anwander A, von Kriegstein K. Altered Structural Connectivity of the Left Visual Thalamus in Developmental Dyslexia. Curr Biol. 2017 Dec 4;27(23):3692-3698.e4. doi: 10.1016/j.cub.2017.10.034. Epub 2017 Nov 16. PMID 29153326
- [Result] Tschentscher N, Ruisinger A, Blank H, Diaz B, von Kriegstein K. Reduced Structural Connectivity Between Left Auditory Thalamus and the Motion-Sensitive Planum Temporale in Developmental Dyslexia. J Neurosci. 2019 Feb 27;39(9):1720-1732. doi: 10.1523/JNEUROSCI.1435-18.2018. Epub 2019 Jan 14. PMID 30643025
- [Result] Kirimoto H, Ogata K, Onishi H, Oyama M, Goto Y, Tobimatsu S. Transcranial direct current stimulation over the motor association cortex induces plastic changes in ipsilateral primary motor and somatosensory cortices. Clin Neurophysiol. 2011 Apr;122(4):777-83. doi: 10.1016/j.clinph.2010.09.025. Epub 2010 Nov 11. PMID 21074492
- [Result] Turkeltaub PE, Benson J, Hamilton RH, Datta A, Bikson M, Coslett HB. Left lateralizing transcranial direct current stimulation improves reading efficiency. Brain Stimul. 2012 Jul;5(3):201-207. doi: 10.1016/j.brs.2011.04.002. Epub 2011 May 5. PMID 22305346
- [Result] Younger JW, Randazzo Wagner M, Booth JR. Weighing the Cost and Benefit of Transcranial Direct Current Stimulation on Different Reading Subskills. Front Neurosci. 2016 Jun 7;10:262. doi: 10.3389/fnins.2016.00262. eCollection 2016. PMID 27375421
- [Result] Younger JW, Booth JR. Parietotemporal Stimulation Affects Acquisition of Novel Grapheme-Phoneme Mappings in Adult Readers. Front Hum Neurosci. 2018 Mar 23;12:109. doi: 10.3389/fnhum.2018.00109. eCollection 2018. PMID 29628882
- [Result] Heth I, Lavidor M. Improved reading measures in adults with dyslexia following transcranial direct current stimulation treatment. Neuropsychologia. 2015 Apr;70:107-13. doi: 10.1016/j.neuropsychologia.2015.02.022. Epub 2015 Feb 19. PMID 25701796
- [Result] Costanzo F, Varuzza C, Rossi S, Sdoia S, Varvara P, Oliveri M, Koch G, Vicari S, Menghini D. Reading changes in children and adolescents with dyslexia after transcranial direct current stimulation. Neuroreport. 2016 Mar 23;27(5):295-300. doi: 10.1097/WNR.0000000000000536. PMID 26848997
- [Result] Costanzo F, Varuzza C, Rossi S, Sdoia S, Varvara P, Oliveri M, Giacomo K, Vicari S, Menghini D. Evidence for reading improvement following tDCS treatment in children and adolescents with Dyslexia. Restor Neurol Neurosci. 2016;34(2):215-26. doi: 10.3233/RNN-150561. PMID 26890096
- [Result] Costanzo F, Rossi S, Varuzza C, Varvara P, Vicari S, Menghini D. Long-lasting improvement following tDCS treatment combined with a training for reading in children and adolescents with dyslexia. Neuropsychologia. 2019 Jul;130:38-43. doi: 10.1016/j.neuropsychologia.2018.03.016. Epub 2018 Mar 14. PMID 29550525
- [Result] Rios DM, Correia Rios M, Bandeira ID, Queiros Campbell F, de Carvalho Vaz D, Lucena R. Impact of Transcranial Direct Current Stimulation on Reading Skills of Children and Adolescents With Dyslexia. Child Neurol Open. 2018 Oct 4;5:2329048X18798255. doi: 10.1177/2329048X18798255. eCollection 2018. PMID 30306098
- [Result] Lazzaro G, Costanzo F, Varuzza C, Rossi S, De Matteis ME, Vicari S, Menghini D. Individual differences modulate the effects of tDCS on reading in children and adolescents with dyslexia. Scientific Studies of Reading. 2021; 25(6): 1-17.
- [Result] Lazzaro G, Costanzo F, Varuzza C, Rossi S, Vicari S, Menghini D. Effects of a short, intensive, multi-session tDCS treatment in developmental dyslexia: Preliminary results of a sham-controlled randomized clinical trial. Prog Brain Res. 2021;264:191-210. doi: 10.1016/bs.pbr.2021.01.015. PMID 34167656
- [Result] Battisti A, Lazzaro G, Costanzo F, Varuzza C, Rossi S, Vicari S, Menghini D. Effects of a short and intensive transcranial direct current stimulation treatment in children and adolescents with developmental dyslexia: A crossover clinical trial. Front Psychol. 2022 Sep 9;13:986242. doi: 10.3389/fpsyg.2022.986242. eCollection 2022. PMID 36160506
- [Derived] Somma F, Lazzaro G, Rima S, Rainich K, Muller-Axt C, Schmid MC, Vicari S, von Kriegstein K, Menghini D. Detecting the contribution of V5/MT in reading, reading-related tasks, eye-movements and EEG-oscillations in children and adolescents with developmental dyslexia via high-definition tDCS: a protocol study. BMC Psychol. 2025 Jul 7;13(1):744. doi: 10.1186/s40359-025-03036-w. PMID 40624571